CLINICAL TRIAL: NCT02944669
Title: Long-Term, Prospective, Non-Interventional Study Monitoring Safety and Training in Patients With Spinal Cord Injuries and Their Trained Companions Recently Initiated With the ReWalk™ Personal Device
Brief Title: ReWalk Personal Device Postmarket Study
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: ReWalk Robotics, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: RW-401
Record Dates: First submitted 2016-10-24; First posted 2016-10-26 (Estimated); Last update posted 2017-02-02 (Estimated); Status verified 2017-02

CONDITIONS: Injuries, Spinal Cord
MeSH Terms: conditions — Spinal Cord Injuries

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Device: Yes

INTERVENTIONS:
Device: ReWalk Personal Device

SUMMARY:
This study seeks to further evaluate the Multi-Tiered Training Program and to further explore the overall safety profile of the ReWalk Personal Device outside of the institutional setting under conditions of routine medical practice.

DETAILED DESCRIPTION:
This study will monitor and further describe the long-term safety of the ReWalk Personal Device for Subjects and their Companions in institutional and non-institutional environments, such as the clinic, home, and community. The study will also evaluate the adequacy of the Multi-Tiered Training Program of the ReWalk Personal Device for Subjects, their Companions, and their Clinical Trainers, monitor and further describe all ReWalk Personal Device malfunctions and screen for potential Unexpected Adverse Events.

ELIGIBILITY:
Inclusion Criteria:

* For use in institutional and non-institutional environments: Subjects with spinal cord injury at levels T7 to L5.
* Age ≥ 18 years old;
* Hands and shoulders can support crutches or a walker;
* Healthy bone density;
* Skeleton does not suffer from any fractures;
* Able to stand using a device such as EasyStand;
* In general good health;
* Height is between 160 cm and 190 cm (5'3" - 6'2");
* Weight does not exceed 100 kg (220 lbs);
* Proficiency in spoken and written English language.

Exclusion Criteria:

* History of severe neurological injuries or disease other than SCI (MS, CP, ALS, TBI, etc.);
* Severe concurrent medical disease, including infections, circulatory, heart or lung, pressure sores;
* Severe spasticity (Ashworth 4)
* Uncontrolled clonus;
* Unstable spine or unhealed limbs or pelvic fractures;
* Heterotopic ossification;
* Significant contractures;
* Psychiatric or cognitive situations that may interfere with proper operation of the device or participation in this study;
* Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Individuals with spinal cord injury at levels T7 to L5 and a prescription for the device.
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2016-06; Primary Completion 2019-09 (Estimated); Study Completion 2019-09 (Estimated)

PRIMARY OUTCOMES:
Long-term safety of the ReWalk Personal Device for Subjects in institutional and non- institutional environments, as measured by 12-month incidence of all Serious Adverse Events in Subjects | 12 Months
Long-term safety of the ReWalk Personal Device for Subjects in institutional and non- institutional environments, as measured by 12-month incidence of falls and fall- associated injuries | 12 Months
Long-term safety of the ReWalk Personal Device for Companions in institutional and non-institutional environments, as measured by 12-month incidence of all Serious Adverse Events in Companions | 12 Months
Adequacy of the Multi-Tiered Training Program of the ReWalk Personal Device for Subjects, as measured by the proportion of Subjects enrolled in training who successfully complete the intended training | 12 Months
Adequacy of the ReWalk Training Program for Subjects, measured by the proportion of Subjects who successfully completed the intended training who are able to demonstrate proficiencies at 12 months after completion of the intended training | 12 Months
Adequacy of the Multi-Tiered Training Program of the ReWalk Personal Device for Subjects, as measured by the Subjects' abilities to navigate surfaces and environments outside of the institutional environment in accordance with their training | 12 Months
Adequacy of the Multi-Tiered Training Program of the ReWalk Personal Device for Companions, as measured by the proportion of Companions enrolled in training who successfully complete the intended training | 12 Months

SECONDARY OUTCOMES:
Reliability of the ReWalk Personal Device, as measured by the rates of all device malfunctions | 12 Months
Adequacy of the Multi-Tiered Training Program of the ReWalk Personal Device for Subjects, as measured by the qualitative Prescribing Physician, Clinical Trainer, Companion, and Subject responses to directed and open-ended questioning | 12 Months
Adequacy of the Multi-Tiered Training Program of the ReWalk Personal Device for Companions, as measured by the qualitative Prescribing Physician, Clinical Trainer, Companion, and Subject responses to directed and open-ended questioning | 12 Months
Adequacy of the Multi-Tiered Training Program of the ReWalk Personal Device for Clinical Trainers, as measured by the qualitative Clinical Trainer responses to directed and open-ended questioning | 12 Months

CONTACTS AND LOCATIONS:
Overall Officials: Mathew Smuck, MD, Principal Investigator — Stanford University
Locations (3):
- United States (3):
  - Stanford University, Palo Alto, California
  - Casa Colina Hospital, Pomona, California
  - Rehabilitation Hospital of Indiana, Indianapolis, Indiana

IPD SHARING:
Plan to Share IPD: Yes
De-identified IPD will be made available after the 3-, 6-, and 12-month intervals.